CLINICAL TRIAL: NCT03964974
Title: Reducing Cannabis Use for Sleep Among Adults Using Medical Cannabis
Acronym: CannSleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark A. Ilgen, Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00151282; 1R34DA047466-01 (NIH)
Record Dates: First submitted 2019-05-17; First posted 2019-05-28 (Actual); Results first posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Insomnia Chronic; Cannabis Use
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy for Insomnia in Cannabis Users (CBTi-CB) (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia in Cannabis Users (CBTi-CB)
- Sleep Hygiene Education (SHE) (Placebo Comparator)
  Interventions: Behavioral: Sleep Hygiene Education (SHE)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia in Cannabis Users (CBTi-CB) — Each CBTi-CB therapy session will review the previous week of sleep/wake diaries and summarize key sleep parameters with participants. The treatment will address cannabis use by increasing use of appropriate coping strategies and improving self-efficacy to manage insomnia and next-day consequences. The content includes: (1) Sleep Scheduling Strategies to consolidate sleep using behavioral strategies that increase the drive for sleep and stabilize the circadian timing system; (2) Sleep Hygiene to discuss behaviors, substances, and environmental conditions that can help or hinder sleep; (3) Cognitive Therapy aims to identify and alter dysfunctional beliefs about sleep and functioning that contribute to insomnia; (4) Counter-Arousal Strategies address ruminative thoughts and increased body tension interfering with ability to fall or return to sleep; (5) Relapse Prevention for Insomnia reviews treatment gains and the behavioral and cognitive strategies that were most helpful.
  Other Names: Cognitive Behavioral Therapy
  Arms: Cognitive Behavioral Therapy for Insomnia in Cannabis Users (CBTi-CB)
Behavioral: Sleep Hygiene Education (SHE) — The SHE condition will be matched to the CBTi-CB condition in terms of level of attention and the non-specific aspects of receiving social support from a study therapist, without providing individualized recommendations. The current content includes: (1) Insomnia History of the participant, including triggers that initiated the problem, duration, severity, and frequency, premorbid sleep characteristics, and previous sleep treatments; (2) Sleep Education about why we sleep, sleep stages, sleep regulation at night, and sleep changes across lifespan; (3) Substance Use and Sleep and the effects of cannabis and other licit and illicit substances on sleep; (4) Environmental Factors that contribute to a sleep-conducive environment; (5) Lifestyle Factors like the effects of diet, exercise, and napping on sleep; (6) Sleep Maintenance Strategies to review treatment gains from the participant's perspective and emphasize the principles covered to maintain sleep improvements.
  Arms: Sleep Hygiene Education (SHE)

SUMMARY:
As medical cannabis use becomes more common in the United States, it is essential to understand the ways in which adults who use medical cannabis perceive the benefits of cannabis use and to identify effective strategies to help them cope with these problems. Emerging data indicate that insomnia and/or use of cannabis for sleep are very common in medical cannabis patients. The present study will adapt and gather pilot data on the impact of a Cognitive Behavioral Therapy for insomnia (CBTi-CB) intervention on sleep- and cannabis-related outcomes in adults who use medical cannabis.

DETAILED DESCRIPTION:
In recent years, the movement to promote the legalization of medical cannabis has grown in the United States and now 29 States and the District of Columbia have provisions that allow for the use of cannabis for medical reasons. Irrespective of the specific reasons for seeking medical cannabis, adults who have been evaluated for medical cannabis certification report significant sleep-related problems as well as frequent use of cannabis to address their sleep problems. Cannabis use for sleep is a key potential target for interventions given that prior research has found that, among individuals with cannabis use disorders, poor sleep is a barrier to sustained remission from cannabis use. Cognitive Behavioral Therapy (CBT) for insomnia is highly effective in individuals with insomnia comorbid with other health conditions, including substance use disorders; however, existing efficacy trials have not specifically evaluated its benefit in those who use cannabis for insomnia. The impact of CBT for insomnia on either sleep or cannabis use in medical cannabis users is, therefore, unknown. The objectives of this project are to adapt and tailor a telephone-delivered CBT for insomnia for adults who use medical cannabis (CBTi-CB) and to evaluate the acceptability and feasibility of this intervention. Qualitative and quantitative data will be collected to refine an existing CBTi-CB protocol and conduct a pilot test of the modified intervention in adults who use medical cannabis. Adults seeking certification for medical cannabis will be approached while waiting for their appointment and screened for insomnia as well as cannabis use for sleep. After initial qualitative interviews and beta testing, eligible participants (N = 60) will be randomized to CBTi-CB or Sleep Hygiene Education (SHE) control condition, delivered over the telephone. Participants will provide self-report data on sleep/insomnia, functioning and cannabis use and objective data on sleep quality will be measured by actigraphy. The study will evaluate changes in self-reported and objectively measured sleep, functioning and frequency/quantity of cannabis use during treatment and over the course of 18-weeks post-baseline. Completion of the study aims will provide all of the elements required for a future fully-powered randomized trial of the longer-term efficacy of CBTi-CB among those with medical cannabis. This line of research would be the first to evaluate a highly effective sleep-focused intervention and determine the effects on sleep-related and non-sleep-related cannabis use in a non-treatment seeking population.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* Insomnia Severity Index (ISI) score greater than 10 (indicating mild insomnia),
* Use of cannabis on average three times a week for the past three months,
* Self-reported use of cannabis to manage insomnia at least once a week over the past month,
* Positive drug screen for Tetrahydrocannabinol (THC),
* Consistent access to a telephone, smart phone, laptop, or tablet

Exclusion Criteria:

* Individuals who do not understand English,
* Individuals judged unable to provide informed consent (e.g. intoxication, mental incompetence),
* Diagnosis or high suspicion of a sleep disorder based on validated self-report questionnaires,
* Self-reported cancer,
* Self-reported pregnancy,
* Self-reported rotating or night (3rd) shift work.
* Participants taking medications for sleep will be included if they meet study criteria for insomnia, medications have been stable for at least 8 weeks, and they agree to maintain the same regimen throughout the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Bloom City Club, Ann Arbor, Michigan
  - Om of Medicine, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnedt JT, Conroy DA, Armitage R, Brower KJ. Cognitive-behavioral therapy for insomnia in alcohol dependent patients: a randomized controlled pilot trial. Behav Res Ther. 2011 Apr;49(4):227-33. doi: 10.1016/j.brat.2011.02.003. Epub 2011 Feb 15. PMID 21377144
- [Background] Ilgen MA, Bohnert K, Kleinberg F, Jannausch M, Bohnert AS, Walton M, Blow FC. Characteristics of adults seeking medical marijuana certification. Drug Alcohol Depend. 2013 Oct 1;132(3):654-9. doi: 10.1016/j.drugalcdep.2013.04.019. Epub 2013 May 15. PMID 23683791
- [Background] Ashrafioun L, Bohnert KM, Jannausch M, Ilgen MA. Characteristics of substance use disorder treatment patients using medical cannabis for pain. Addict Behav. 2015 Mar;42:185-8. doi: 10.1016/j.addbeh.2014.11.024. Epub 2014 Nov 26. PMID 25481452
- [Background] Cranford JA, Arnedt JT, Conroy DA, Bohnert KM, Bourque C, Blow FC, Ilgen M. Prevalence and correlates of sleep-related problems in adults receiving medical cannabis for chronic pain. Drug Alcohol Depend. 2017 Nov 1;180:227-233. doi: 10.1016/j.drugalcdep.2017.08.017. Epub 2017 Sep 9. PMID 28926791
- [Background] Arnedt JT, Cuddihy L, Swanson LM, Pickett S, Aikens J, Chervin RD. Randomized controlled trial of telephone-delivered cognitive behavioral therapy for chronic insomnia. Sleep. 2013 Mar 1;36(3):353-62. doi: 10.5665/sleep.2448. PMID 23450712
- See also: SAMHSA National Survey on Drug Use and Health data — https://www.samhsa.gov/data/data-we-collect/nsduh-national-survey-drug-use-and-health
- See also: Medical Marijuana laws by state — http://www.ncsl.org/research/health/state-medical-marijuana-laws.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Behavioral Therapy for Insomnia in Cannabis Users (CBTi-CB): Each CBTi-CB therapy session reviewed the previous week of sleep/wake diaries and summarize key sleep parameters with participants. The treatment addressed cannabis use by increasing use of appropriate coping strategies and improving self-efficacy to manage insomnia and next-day consequences. The content includes: (1) Sleep Scheduling Strategies to consolidate sleep using behavioral strategies that increase the drive for sleep and stabilize the circadian timing system; (2) Sleep Hygiene to discuss behaviors, substances, and environmental conditions that can help or hinder sleep; (3) Cognitive Therapy aims to identify and alter dysfunctional beliefs about sleep and functioning that contribute to insomnia; (4) Counter-Arousal Strategies address ruminative thoughts and increased body tension interfering with ability to fall or return to sleep; (5) Relapse Prevention for Insomnia reviews treatment gains and the behavioral and cognitive strategies that were most helpful.
- Sleep Hygiene Education (SHE): The SHE condition was matched to the CBTi-CB condition in terms of level of attention and the non-specific aspects of receiving social support from a study therapist, without providing individualized recommendations. The current content includes: (1) Insomnia History of the participant, including triggers that initiated the problem, duration, severity, and frequency, premorbid sleep characteristics, and previous sleep treatments; (2) Sleep Education about why we sleep, sleep stages, sleep regulation at night, and sleep changes across lifespan; (3) Substance Use and Sleep and the effects of cannabis and other licit and illicit substances on sleep; (4) Environmental Factors that contribute to a sleep-conducive environment; (5) Lifestyle Factors like the effects of diet, exercise, and napping on sleep; (6) Sleep Maintenance Strategies to review treatment gains from the participant's perspective and emphasize the principles covered to maintain sleep improvements.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy for Insomnia in Cannabis Users (CBTi-CB) | Sleep Hygiene Education (SHE)
Started | 30 | 27
Assigned and Received Intervention | 26 | 21
8 Week Follow Up | 26 | 22
16 Week Follow Up | 27 | 22
Completed | 27 | 22
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- CBTi-CB: Cognitive Behavioral Therapy for Insomnia in Cannabis Users
  Cognitive Behavioral Therapy for Insomnia in Cannabis Users: Each CBTi-CB therapy session reviewed the previous week of sleep/wake diaries and summarize key sleep parameters with participants. The treatment addressed cannabis use by increasing use of appropriate coping strategies and improving self-efficacy to manage insomnia and next-day consequences. The content includes: (1) Sleep Scheduling Strategies to consolidate sleep using behavioral strategies that increase the drive for sleep and stabilize the circadian timing system; (2) Sleep Hygiene to discuss behaviors, substances, and environmental conditions that can help or hinder sleep; (3) Cognitive Therapy aims to identify and alter dysfunctional beliefs about sleep and functioning that contribute to insomnia; (4) Counter-Arousal Strategies address ruminative thoughts and increased body tension interfering with ability to fall or return to sleep; (5) Relapse Prevention for Insomnia reviews treatment gains and the behavioral and cognitive strategies that were most helpful.
- Sleep Hygiene Education: Sleep Hygiene Education
  The SHE condition was matched to the CBTi-CB condition in terms of level of attention and the non-specific aspects of receiving social support from a study therapist, without providing individualized recommendations. The current content includes: (1) Insomnia History of the participant, including triggers that initiated the problem, duration, severity, and frequency, premorbid sleep characteristics, and previous sleep treatments; (2) Sleep Education about why we sleep, sleep stages, sleep regulation at night, and sleep changes across lifespan; (3) Substance Use and Sleep and the effects of cannabis and other licit and illicit substances on sleep; (4) Environmental Factors that contribute to a sleep-conducive environment; (5) Lifestyle Factors like the effects of diet, exercise, and napping on sleep; (6) Sleep Maintenance Strategies to review treatment gains from the participant's perspective and emphasize the principles covered to maintain sleep improvements.
- Total: Total of all reporting groups
Arm/Group | CBTi-CB | Sleep Hygiene Education | Total
Number analyzed (Participants) | 30 | 27 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (12.0) | 38.7 (13.7) | 37.6 (12.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 7 | 7 | 14
  Non-Binary | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 30 | 25 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 24 | 23 | 47
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 27 | 57
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: units on a scale] — The range of the ISI is 0 to 28, with 28 corresponding to maximum severity.
  units on a scale | 17.4 (4.5) | 16.2 (3.8) | 16.8 (4.2)
Frequency of Cannabis Use [Count of Participants; unit: Participants]
  Participants Who Used 2 - 3 Times/Week | 4 | 3 | 7
  Participants Who Used 4 or More Times/Week | 26 | 24 | 50
Cannabis Use Per Day [Count of Participants; unit: Participants]
  Less Than Daily Use | 2 | 1 | 3
  1 - 2 Times Per Day | 10 | 12 | 22
  3 - 4 Times Per Day | 15 | 10 | 25
  5 or More Times Per Day | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Insomnia Severity Index Score at Study Completion
Description: The Insomnia Severity Index (ISI) is a brief self-report instrument measuring the patient's perception of both nocturnal and diurnal symptoms of insomnia.
  The ISI comprises seven items assessing the perceived severity of difficulties initiating sleep, staying asleep, and early morning awakenings, satisfaction with current sleep pattern, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. The range of the ISI is 0 to 28, with 28 corresponding to maximum severity.
Time Frame: 16 Weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Cognitive Behavioral Therapy for Insomnia in Cannabis Users (CBTi-CB): Each CBTi-CB therapy session reviewed the previous week of sleep/wake diaries and summarized key sleep parameters with participants. The treatment addressed cannabis use by increasing use of appropriate coping strategies and improving self-efficacy to manage insomnia and next-day consequences. The content included: (1) Sleep Scheduling Strategies to consolidate sleep using behavioral strategies that increase the drive for sleep and stabilize the circadian timing system; (2) Sleep Hygiene to discuss behaviors, substances, and environmental conditions that can help or hinder sleep; (3) Cognitive Therapy aims to identify and alter dysfunctional beliefs about sleep and functioning that contribute to insomnia; (4) Counter-Arousal Strategies address ruminative thoughts and increased body tension interfering with ability to fall or return to sleep; (5) Relapse Prevention for Insomnia reviews treatment gains and the behavioral and cognitive strategies that were most helpful.
- Sleep Hygiene Education (SHE): The SHE condition was matched to the CBTi-CB condition in terms of level of attention and the non-specific aspects of receiving social support from a study therapist, without providing individualized recommendations. The content included: (1) Insomnia History of the participant, including triggers that initiated the problem, duration, severity, and frequency, premorbid sleep characteristics, and previous sleep treatments; (2) Sleep Education about why we sleep, sleep stages, sleep regulation at night, and sleep changes across lifespan; (3) Substance Use and Sleep and the effects of cannabis and other licit and illicit substances on sleep; (4) Environmental Factors that contribute to a sleep-conducive environment; (5) Lifestyle Factors like the effects of diet, exercise, and napping on sleep; (6) Sleep Maintenance Strategies to review treatment gains from the participant's perspective and emphasize the principles covered to maintain sleep improvements.
Arm/Group | Cognitive Behavioral Therapy for Insomnia in Cannabis Users (CBTi-CB) | Sleep Hygiene Education (SHE)
Number analyzed (Participants) | 30 | 27
units on a scale
  Longitudinal Model estimates at 8-week Follow-up | 11.2 (0.8) | 12.6 (0.8)
  Longitudinal Model estimates at 16-week Follow-up | 6.0 (1.1) | 8.8 (1.0)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy for Insomnia in Cannabis Users (CBTi-CB) vs Sleep Hygiene Education (SHE); Persons in the CBTI-CB condition were hypothesized as realizing greater reduction in insomnia severity as measured by the Insomnia Severity Index (ISI) over time compared to the Sleep Hygiene Education (SHE) condition. 80% power was estimated to detect a medium or larger effect size (d>0.52) on sleep- and functioning-related outcomes, even with a more conservative alpha set at 0.017 (i.e., 0.05/3 for the 3 outcomes); Test type: Superiority — 2-sided hypothesis tests were utilized to compare ISI score over time in the two treatment conditions; p = 0.0041, Mixed Models Analysis — This is the calculated p-value. The threshold for statistical significance was 0.05; Median Difference (Final Values) = -4.307, 95% CI 2-sided [-7.510 to -1.104], Standard Error of Mean 1.612; Parameter is estimated difference in final means, CBTi-CB - Control. Minus sign denotes greater decrease for CBTi-CB. Effect size for Time X Condition = 0.81

ADVERSE EVENTS:
Time Frame: 16 Weeks
Groups:
- Sleep Education: Psycho-education on sleep and sleep hygiene
  Sleep Education: The SE condition was matched to the CBTi-CB condition in terms of level of attention and the non-specific aspects of receiving social support from a study therapist, without providing individualized recommendations. The current content includes: (1) Insomnia History of the participant, including triggers that initiated the problem, duration, severity, and frequency, premorbid sleep characteristics, and previous sleep treatments; (2) Sleep Education about why we sleep, sleep stages, sleep regulation at night, and sleep changes across lifespan; (3) Substance Use and Sleep and the effects of cannabis and other licit and illicit substances on sleep; (4) Environmental Factors that contribute to a sleep-conducive environment; (5) Lifestyle Factors like the effects of diet, exercise, and napping on sleep; (6) Sleep Maintenance Strategies to review treatment gains from the participant's perspective and emphasize the principles covered to maintain sleep improvements.
Arm/Group | CBTi-CB | Sleep Education
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/27
Other Adverse Events (participants affected / at risk) | 0/30 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT03964974/Prot_SAP_001.pdf
  • Informed Consent Form (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT03964974/ICF_000.pdf